CLINICAL TRIAL: NCT02792673
Title: Comparative Study Between Three Different Embryo Transfer Media: Hyaluronan-enriched Medium "Embryo Glue®", 30% Protein-supplemented Culture Medium "Global Total®" and Autologous Follicular Fluid Concerning "Chemical and Clinical" Pregnancy Rate and "Ongoing Pregnancy and Miscarriage" Rates in ICSI Cycles
Brief Title: Comparative Study of Three Different Embryo Transfer Media in ICSI Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Collaborators: Ibn Sina Hospital (Other Government); Qena Fertility Center, Qena, Egypt (Unknown)
Responsible Party: Principal Investigator, Ahmed Mowafy, Investigator, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Assisted Reproduction Unit - 1
Record Dates: First submitted 2016-05-23; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Improvement of Embryo Transfer Technique; Improvement of Implantation
Keywords: Embryo transfer media; improvement of embryo transfer technique; improvement of implantation; Hyaluronan-enriched media "Embryo Glue®"; 30% Protein-supplemented Culture Medium "Global Total®"; Autologous Follicular Fluid as embryo transfer medium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- "Embryo Glue®" (Active Comparator): Hyaluronan-enriched medium
  Interventions: Other: embryos will be transferred using a medium of 0.5 mg/mL of Hyaluronan-enriched medium (EmbryoGlue®, Vitrolife, Sweden); Device: Labotect embryo transfer catheter
- "Global Total®" (Active Comparator): 30% Protein-supplemented Culture Medium
  Interventions: Other: embryos will be transferred using a medium of 30% Protein-supplemented Culture Medium (Global total®, Life Global group, Canada); Device: Labotect embryo transfer catheter
- Autologous Follicular Fluid (Experimental): a novel technique
  Interventions: Other: a novel technique in which embryos will be transferred using a medium of autologous Follicular Fluid; Device: Labotect embryo transfer catheter

INTERVENTIONS:
Other: embryos will be transferred using a medium of 0.5 mg/mL of Hyaluronan-enriched medium (EmbryoGlue®, Vitrolife, Sweden)
  Arms: "Embryo Glue®"
Other: embryos will be transferred using a medium of 30% Protein-supplemented Culture Medium (Global total®, Life Global group, Canada)
  Arms: "Global Total®"
Other: a novel technique in which embryos will be transferred using a medium of autologous Follicular Fluid
  Arms: Autologous Follicular Fluid
Device: Labotect embryo transfer catheter

SUMMARY:
The study design is a prospective randomized uncontrolled clinical trial. It will include 150 cases.

The aim of this study is to compare the efficacy of three different media used for embryo transfer regarding "chemical and clinical" pregnancy rate, implantation rate and ongoing pregnancy and miscarriage rates in IVF and ICSI cycles.

The three different embryo transfer media are:

1. Hyaluronan-enriched medium "Embryo Glue®"
2. 30% Protein-supplemented Culture medium "Global Total®"
3. Autologous Follicular Fluid (a Novel technique) In order to establish the optimal media for embryo transfer

DETAILED DESCRIPTION:
Two or three embryos will be transferred at day 5 after ovum pick-up (OPU).

The patients will be divided randomly (closed envelop method) into 3 groups:

* Group A (50 patients): embryos will be transferred using a medium supplemented with 0.5 mg/mL of hyaluronic acid (EmbryoGlue®, Vitrolife, Sweden) for 20 minutes before intrauterine transfer took place
* Group B (50 patients): embryos will be transferred using a medium of 30% Protein-supplemented Culture Medium (Global total®, Life Global group, Canada) for 20 minutes.
* Group C (50 patients): a novel technique in which embryos will be transferred using a medium of autologous Follicular Fluid for 20 minutes.

Follicular fluid will be collected in a sterile procedure, centrifuged for 20 minutes in an embryo test tube. The supernatant will be removed in a sterilized technique then heated to 56°C for 30 minutes then filtered through 0.22 micron filter. Gentamycin sulphate will be added at a concentration of 10 µg/mL then the liquid is preserved in a normal freezer.

Defreezing follicular fluid will be performed at day-1 before embryo transfer. The follicular fluid will be warmed to room temperature. Preparation of embryo transfer media will be performed as usual, will be covered with paraffin oil (Ovoil®, Vitrolife, Sweeden) and then incubated overnight in 7% CO2, 9% O2, 22% N2.

All embryo transfers will be performed using an embryo transfer catheter (Labotect catheter, Labotect GmbH, Germany).

Number of embryos transferred will be according to ASRM guideline 2013 on day 5 after ovum pick-up (OPU).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-35 years
2. Body mass index (BMI): ≤ 30
3. Anti-mullerian hormone (AMH): 1.1 - 3
4. No gynecological problem e.g. fibroid, endometriosis, uterine polyp, hydrosalpinx or adenomysis
5. Male factor: mild to moderate oligo or asthenospermia

Exclusion Criteria:

1. Age: <18 years or >35 years
2. Body mass index (BMI): >30
3. Anti-mullerian hormone (AMH): <1.1 or >3
4. gynecological problem e.g. fibroid, endometriosis, uterine polyp, hydrosalpinx or adenomysis will be excluded
5. Male factor: Abnormal sperm morphology; (globozoospermia and pin-point sperm) and azoospermia; (whether obstructive or non-obstructive) will be excluded
6. Patients with recurrent implantation failure

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Chemical pregnancy rate | 14 days after embryo transfer
  assessed by quantitative β hCG in the serum

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6th week of gestation
  assessed by ultrasonic visualization of intrauterine gestational sac

OTHER OUTCOMES:
Implantation rate. | 6th week of gestation
Ongoing pregnancy and miscarriage rates | 12th week of gestation

IPD SHARING:
Plan to Share IPD: Undecided